CLINICAL TRIAL: NCT04903145
Title: Proof-of-concept of the Measurement of Lung Function Using the Relaxed Expiratory Occlusion Monitor (REOM)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Thorasys Thoracic Medical Systems Inc. (Industry)
Collaborators: MedTeq (Industry)
Responsible Party: Sponsor
Other Study IDs: REOM 2019-2053
Record Dates: First submitted 2021-05-19; First posted 2021-05-26 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Asthma in Children
Keywords: tremoflo; oscillometry; interrupter; asthma; REOM
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: REOM — To compare data generated by the REOM device with data from the tremoflo C-100 device

SUMMARY:
(i) To validate the inversed occlusion technique by comparing the results of resistance obtained on the relaxed expiratory occlusion monitor (REOM) with the resistance obtained with respiratory oscillometry (OSC) measurements on the tremoflo® C-100 and (ii) explore (within-test and day-to-day) repeatability and responsiveness to change of this technique when used as home monitoring device in children with asthma.

DETAILED DESCRIPTION:
Children will be evaluated for eligibility by telephone or videoconferencing. After eligibility and consent documented by email by parents and on a source document by the research assistant:

1. Children will receive by courier one new REOM unit, a tablet with charger, and related disposables (nose clips etc.),
2. At a videoconference planned at a mutually conveniently time with the child and their parents the following will be obtained;

   1. Basic demographics (date of birth, age, sex, ethnicity, height, weight) and asthma morbidity and medications.
   2. Training on the REOM unit measurement using a recorded instructions video, followed by hand-on use of the unit under remote observation. The Research Assistant will teach the parents and child in the REOM, namely on how to use the unit to measure resistance until it is mastered and reproducible, how to complete the brief daily questionnaire, and how upload data from the REOM to the tablet by Bluetooth. Confirmation of the validity and reproducibility of the technique will be obtained by review of the measurement output that will be sent by WIFI automatically from the tablet to a protected google drive (with the patient identified only by a code) accessible to the Coordinating Centre.
   3. Briefly, a minimum of three (3) reproducible measurements of Reo on the REOM will be obtained in accordance to the following standardized procedures: the subjects will be asked to be comfortably seated upright, with the head slightly tilted upward at an angle of about 15 degrees from neutral position to prevent upper airway obstruction, with the cheeks tightly supported to prevent upper airway shunting. A nose clip will be worn to prevent nasal air leak. Subjects will be instructed to breathe normally in a single-use bacterial/viral respiratory filter connected to the mouthpiece of the REOM device. This manoeuvre will be repeated for a maximum of 6 trials to obtain a coefficient of variation (CV) ≤15% on at least 3 Reo measurements with visual remote inspection of the curves and results via Bluetooth connection by the research assistant. Each trial will last 20 to 30 seconds to obtain a minimum of 3 to 6 valid expirations per trial. The mean Reo of 3 reproducible measurements will be calculated at the peak (Reo1) and the low (Reo2) flow.
3. Once the technique is mastered, the child will be asked to:

   1. Perform the REOM measurements once daily before receiving their asthma controller medication, ideally at the same time in the evening.
   2. If the child requires a rapid beta-2 agonists because of symptoms, a before and after measurement will be obtained 30 minutes after the dose has been administered to document responsiveness to change once a day when sick.
   3. Once a week, a short questionnaire including the cACT (or ACT for 12 years and older), a question about an acute care visit or use of rescue oral corticosteroids, and occurrence of any adverse event will be sent by text message or email (patient preference) throughout the study duration.
4. A research assistant will contact the family at 7±3 days, 14±3 days, and monthly thereafter or, if in case of problem with the equipment or interruption in REOM measurements/response to the weekly questionnaire.

The study duration will be 4 months (to maximize the chance of an exacerbation).

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 6 and 17 years old
2. Adequate understanding of French or English
3. Asthma diagnosis confirmed by a physician
4. Poor asthma control in the past 6 months, that is,

   1. an acute exacerbation requiring oral corticosteroids, or
   2. an FEV1 <80% of predicted, FEV1/FVC ratio below the lower limit of normal, or significant (≥12%) reversibility in FEV1, or
   3. a total score <20 on the child Asthma Control Test (ACT) for children aged ≤11 years or on the ACT for those aged ≥12 years).

Exclusion Criteria:

1. Inability to produce a good seal around the mouthpiece when previously tested with spirometry
2. Oscillometry or REOM, contra-indication to performing respiratory tests (e.g., facial trauma, chest pain, severe scoliosis)
3. Other reason interfering with respiratory testing.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The asthmatic study subjects will be recruited a the Sainte-Justine University Hospital Center, Montreal, QC. Recruitment will be performed by Dr. Ducharme's research staff. The study will be conducted remotely with patients who consented to the Pediatric asthma database and Biobank of the Sainte-Justine University Hospital Center or among the families subscribing to the Asthma Clinic newsletter or seeing the advertisement on the CHUSJ website.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Respiratory resistance R5 | Over one week
  Using the tremoflo C-100 at 5 Hz to calculate the mean resistance during the patient's tidal breathing.
Expiratory resistance (R5exp) | Over one week
  Using the tremoflo C-100 at 5 Hz to calculate resistance during the patient's exhalation.
Resistance at low expiratory flow (Reo2) | Over one week
  Using the REOM device the resistance (Reo2) at low expiratory flow will be calculated.

SECONDARY OUTCOMES:
Respiratory resistance R19 | Over one week
  Using the tremoflo C-100 at 19 Hz to calculate the mean resistance during the patient's tidal breathing.
Expiratory resistance (R19exp) | Over one week
  Using the tremoflo C-100 at 19 Hz to calculate resistance during the patient's exhalation.
Resistance at high expiratory flow (Reo1) | Over one week
  Using the REOM device the resistance (Reo1) at high expiratory flow will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Francine M Ducharme, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- Sainte-Justine University Hospital Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaminsky DA. What does airway resistance tell us about lung function? Respir Care. 2012 Jan;57(1):85-96; discussion 96-9. doi: 10.4187/respcare.01411. PMID 22222128
- [Background] Lamontagne AJ, Pelaez S, Grad R, Blais L, Lavoie KL, Bacon SL, Guay H, Gauthier A, McKinney ML, Ernst P, Collin J, Ducharme FM. Facilitators and solutions for practicing optimal guided asthma self-management: the physician perspective. Can Respir J. 2013 Jul-Aug;20(4):285-93. doi: 10.1155/2013/146839. PMID 23936888
- [Background] Kaplan A, Stanbrook M. Must family physicians use spirometry in managing asthma patients?: YES. Can Fam Physician. 2010 Feb;56(2):126, 128, 130,132; discussion e49, e51. No abstract available. PMID 20154239
- [Background] Lundblad LKA, Blouin N, Grudin O, Grudina L, Drapeau G, Restrepo N, Ducharme FM. Comparing lung oscillometry with a novel, portable flow interrupter device to measure lung mechanics. J Appl Physiol (1985). 2021 Apr 1;130(4):933-940. doi: 10.1152/japplphysiol.01072.2020. Epub 2021 Feb 4. PMID 33539262
- [Background] Lougheed MD, Lemiere C, Ducharme FM, Licskai C, Dell SD, Rowe BH, Fitzgerald M, Leigh R, Watson W, Boulet LP; Canadian Thoracic Society Asthma Clinical Assembly. Canadian Thoracic Society 2012 guideline update: diagnosis and management of asthma in preschoolers, children and adults. Can Respir J. 2012 Mar-Apr;19(2):127-64. doi: 10.1155/2012/635624. PMID 22536582
- [Background] Bates JH, Irvin CG, Farre R, Hantos Z. Oscillation mechanics of the respiratory system. Compr Physiol. 2011 Jul;1(3):1233-72. doi: 10.1002/cphy.c100058. PMID 23733641
- [Background] Goldman MD, Saadeh C, Ross D. Clinical applications of forced oscillation to assess peripheral airway function. Respir Physiol Neurobiol. 2005 Aug 25;148(1-2):179-94. doi: 10.1016/j.resp.2005.05.026. PMID 15990365
- [Background] MEAD J, WHITTENBERGER JL. Evaluation of airway interruption technique as a method for measuring pulmonary airflow resistance. J Appl Physiol. 1954 Jan;6(7):408-16. doi: 10.1152/jappl.1954.6.7.408. No abstract available. PMID 13117773
- [Background] Ducharme FM, Jroundi I, Jean G, Lavoie Boutin G, Lawson C, Vinet B. Interdevice agreement in respiratory resistance values by oscillometry in asthmatic children. ERJ Open Res. 2019 Mar 18;5(1):00138-2018. doi: 10.1183/23120541.00138-2018. eCollection 2019 Feb. PMID 30895187
- [Background] Oostveen E, MacLeod D, Lorino H, Farre R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003 Dec;22(6):1026-41. doi: 10.1183/09031936.03.00089403. PMID 14680096
- [Background] Jones SR, Carley S, Harrison M. An introduction to power and sample size estimation. Emerg Med J. 2003 Sep;20(5):453-8. doi: 10.1136/emj.20.5.453. PMID 12954688
- [Background] Shi Y, Aledia AS, Tatavoosian AV, Vijayalakshmi S, Galant SP, George SC. Relating small airways to asthma control by using impulse oscillometry in children. J Allergy Clin Immunol. 2012 Mar;129(3):671-8. doi: 10.1016/j.jaci.2011.11.002. Epub 2011 Dec 17. PMID 22178635
- [Background] Robinson PD, Brown NJ, Turner M, Van Asperen P, Selvadurai H, King GG. Increased day-to-day variability of forced oscillatory resistance in poorly controlled or persistent pediatric asthma. Chest. 2014 Oct;146(4):974-981. doi: 10.1378/chest.14-0288. PMID 24991854
- [Background] Wong A, Hardaker K, Field P, Huvanandana J, King GG, Reddel H, Selvadurai H, Thamrin C, Robinson PD. Home-based Forced Oscillation Technique Day-to-Day Variability in Pediatric Asthma. Am J Respir Crit Care Med. 2019 May 1;199(9):1156-1160. doi: 10.1164/rccm.201809-1659LE. No abstract available. PMID 30822109
- [Background] Guyatt GH, Kirshner B, Jaeschke R. Measuring health status: what are the necessary measurement properties? J Clin Epidemiol. 1992 Dec;45(12):1341-5. doi: 10.1016/0895-4356(92)90194-r. PMID 1460470